CLINICAL TRIAL: NCT02525471
Title: A Pilot Study of RNS60 in Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sabrina Paganoni, M.D. (Other)
Responsible Party: Sponsor-Investigator, Sabrina Paganoni, M.D., Principal Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RNS60-01
Record Dates: First submitted 2015-08-12; First posted 2015-08-17 (Estimated); Results first posted 2021-03-03 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: ALS
MeSH Terms: interventions — RNS60; Sodium Chloride; Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RNS60 (Experimental): Following screening visit to determine eligibility, enrolled subjects will undergo the baseline visit within 6 weeks where the first intravenous (IV) infusion of study medication, RNS60, will be administered. Study medication for inhalation use will be dispensed at this time, and again at weeks 7 and 15. Subjects will continue once a week follow ups to receive RNS60 by IV infusion, continuing inhalation use the remaining 6 days per week, for 23 weeks total. Additionally, eligible subjects will undergo PET imaging at baseline and again between weeks 18 and 23.
  In addition, upon nearing completion of the core study, subjects will be given the option to continue to receive drug for approximately an additional 24 weeks, for a total of approximately 48 weeks on study drug, following the optional extension phase schedule of activities.
  Interventions: Drug: RNS60

INTERVENTIONS:
Drug: RNS60 — RNS60 will be administered in two ways: by intravenous (IV) infusion one day a week (infusion dose: 375ml, infused over a 40-min period) and by inhalation (the remaining 6 days a week, 4 ml/day) for 23 weeks.
  In addition, subjects will be given the option to continue to receive drug for approximately an additional 24 weeks, for a total of approximately 48 weeks on study drug. Study drug will be given by intravenous (IV) infusion one day a week (infusion dose: 375ml, infused over a 40-min period) and by inhalation (the remaining 6 days a week, 4 ml/day) during the extension phase.
  Other Names: Electrokinetically Processed Fluid; saline and oxygen

SUMMARY:
The purpose of this study is to determine the safety and tolerability of RNS60 in patients with Amyotrophic lateral sclerosis (ALS). Investigators will also measure the impact of RNS60 on several markers of neuro-inflammation, measured by blood biomarkers and positron emission tomography (PET) imaging.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a fatal, neurodegenerative disease for which there is no cure. A substantial body of evidence implicates the neuroimmune system in ALS pathophysiology. Of relevance to this study, microglia activation in the brain has been found to correlate positively with faster rate of disease progression. In addition, studies of blood cells in people with ALS have shown an increased activation of two of the major inflammatory cell types in the body, monocytes and T cells. Among T cells, regulatory T cells (Tregs) have been recently proposed to play a role in ALS progression.

RNS60 is an electrokinetically altered aqueous fluid. Chemically, RNS60 is composed of saline and oxygen. The electrokinetic processing of RNS60 in Revalesio's patented Revalesio Pump (RP) produces charge-stabilized nanostructures (CSNs) that exhibit electrical fields. RNS60 is available for intravenous administration and inhalation. RNS60 has been extensively tested in preclinical toxicological studies and has shown very little to no side effects. In addition, RNS60 was well tolerated in three phase I human safety studies, one after intravenous administration and two after inhalation.

Preclinical in vitro and in vivo studies in multiple disease models have demonstrated that RNS60 has broad anti-inflammatory effects. These effects include reduction of microglia activation, increase of the Tregs subpopulation of lymphocytes, and neuroprotection in several disease models.

ELIGIBILITY:
Inclusion Criteria:

* Amyotrophic Lateral Sclerosis (ALS) volunteers must be diagnosed as having possible, probable, probable-laboratory supported, or definite ALS, either sporadic or familial according to modified El Escorial criteria.
* Age 18-80, able to provide informed consent, and comply with study procedures.
* Participants must not have taken riluzole for at least 30 days, or be on a stable dose of riluzole for at least 30 days, prior to screening (riluzole-naïve participants are permitted in the study).
* Women must not be able to become pregnant (e.g. post menopausal, surgically sterile, or using adequate birth control) for the duration of the study and 3 months after study completion.
* Males should practice contraception for the duration of the study and 3 months after completion.
* Ability to safely lie flat for 90 min for Positron Emission Tomography (PET) procedures in the opinion of the study physician.
* High or mixed affinity to bind translocator (TSPO) protein (Ala/Ala or Ala/Thr)

Exclusion Criteria:

* Abnormal liver function defined as aspartate aminotransferase (AST) and/or alanine transaminase (ALT) > 3 times the upper limit of the normal.
* Renal insufficiency as defined by a serum creatinine > 1.5 times the upper limit of normal.
* The presence of unstable psychiatric disease, cognitive impairment, or dementia that would impair ability of the participant to provide informed consent, according to PI judgment.
* Clinically significant unstable medical condition (other than ALS) that would pose a risk to the participant if they were to participate in the study.
* History of HIV, clinically significant chronic hepatitis, or other active infection.
* Females must not be lactating or pregnant.
* Active participation in another ALS clinical trial within 30 days of the Screening Visit
* Exposure to immunomodulatory medications within 30 days of the Screening Visit.
* Any contraindication to undergo MRI studies such as

  * History of a cardiac pacemaker or pacemaker wires
  * Metallic particles in the body
  * Vascular clips in the head
  * Prosthetic heart valves
  * Claustrophobia
* Radiation exposure that exceeds the site's current guidelines
* Current use of tobacco products including cigarettes, cigars, snuff and chewing tobacco, or nicotine replacement products such as gum or patch

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-10; Primary Completion 2017-06-21 (Actual); Study Completion 2017-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Paganoni, MD, Principal Investigator — Massachusetts General Hospital; Nazem Atassi, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- RNS60: RNS60 will be administered in two ways: by intravenous (IV) infusion one day a week (infusion dose: 375ml, infused over a 40-min period) and by inhalation (the remaining 6 days a week, 4 ml/day) for 24 weeks.
Period: Overall Study
Arm/Group | RNS60
Started | 24
Randomized/Treated | 16
Completed | 13
Not Completed | 11
Not completed — Screen Failure | 6
Not completed — Withdrawal by Subject | 4
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Although 24 patients signed consent, only 16 patients were treated. Baseline characteristics are reported for these 16 treated patients.
Arm/Group | RNS60
Number analyzed (Participants) | 16
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 52.9 [24.5 to 69.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 16
Disease Onset [Count of Participants; unit: Participants]
  Bulbar onset | 3
  Limb onset | 12
  Other onset | 1
Slow Vital Capacity [Mean (Inter-Quartile Range); unit: Max % predicted] | 63.8 [28.0 to 99.0]
ALS Functional Rating Scale - Revised [Mean (Inter-Quartile Range); unit: units on a scale] — The ALSFRS-R is a quickly administered (5 minute) ordinal rating scale used to determine a subject's assessment of their capability and independence in 12 functional activities. There are 12 questions, graded by the subject 0-4 (4 is normal). Score of 0 (worst) to 48 (best). Reflects speech and swallowing, fine motor skills, large motor skills, and breathing.
  units on a scale | 34.1 [23.0 to 44.0]
Riluzole Use [Count of Participants; unit: Participants] | 16
Months Since Symptom Onset [Mean (Inter-Quartile Range); unit: months] | 30.3 [7.1 to 68.4]

OUTCOME MEASURES:

1. Primary Outcome: Safety as Measured by the Number of Participants Experiencing Adverse Events
Description: Safety will be assessed by the occurrence of adverse events over the course of 24 weeks of treatment plus the 4 week off-drug follow-up period (total of 28 weeks). Per the protocol, the first treatment was administered at Baseline (Day 0) and the 24th treatment was administered at Week 23 (Day 161), and a safety phone call performed at Week 28 (Day 196).
Time Frame: 28 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | RNS60
Number analyzed (Participants) | 16
Participants | 16

2. Primary Outcome: Tolerability to Complete the Entire 24 Week Study on Study Drug
Description: Tolerability will be defined as the ability of subjects to complete the entire 24-week study on study drug. Per the protocol, the first treatment was administered on Day 0 (Baseline) and the 24th treatment was administered at Week 23.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Groups:
- RNS60: RNS60: RNS60 will be administered in two ways: by intravenous (IV) infusion one day a week (infusion dose: 375ml, infused over a 40-min period) and by inhalation (the remaining 6 days a week, 4 ml/day) for 24 weeks.
Arm/Group | RNS60
Number analyzed (Participants) | 16
Participants | 13

3. Primary Outcome: Blood Biomarkers of Inflammation.
Description: Selected biomarkers of inflammation were measured at Baseline and Week 23 on a sub-set of subjects. Biomarkers included IL-17 plasma levels and FOXP3 mRNA expression in whole blood, a marker of Treg function. Per the protocol, the first treatment was administered on Day 0 (Baseline) and the 24th treatment was administered on Day 161 (Week 23).
Time Frame: 24 Weeks
Population: Eleven (11) subjects participated in the imaging sub-study. Blood biomarkers were collected in a selected subset of subjects per protocol inclusion and exclusion criteria. Samples not collected were due to tech difficulties.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | RNS60
Number analyzed (Participants) | 11
pg/ml
  IL-17 change at Week 24: number analyzed (Participants) | 10
  IL-17 change at Week 24 | -25.4 (22.33)
  FOXP3 change at Week 24: number analyzed (Participants) | 8
  FOXP3 change at Week 24 | -0.02 (0.338)

4. Primary Outcome: Change From Baseline in Standardized Uptake Value (SUV) Normalized to Whole Brain Mean (SUVR) at Approximately 60-90 Minutes Post Injection
Description: Glial activation was estimated in a subset of participants by magnetic resonance positron emission tomography (MR-PET) using the [11C]-PBR28 ligand. The subset excludes individuals homozygous for the T/T allele of the Ala147Thr TSPO polymorphism (rs6971) associated with low affinity for [11C]-PBR28. Glial activation was quantified as a mean standardized uptake value (SUV) using PET images acquired 60 to 90 minutes post-injection of approximately 430 MBq [11C]-PBR28. FreeSurfer v6.0 (https://surfer.nmr.mgh.harvard.edu) was employed to circumscribe a region of interest (ROI) defined anatomically as the precentral gyrus and the anterior portion of the paracentral lobule, bilaterally. SUV of the ROI was normalized to the SUV of the whole brain and expressed as a SUV ratio (SUVR) to control for inter-individual variability in the global [11C]-PBR28 PET signal. Per the protocol, the first treatment was administered on Day 0 (Baseline) and the 24th treatment was administered on Day 161 (
Time Frame: 24 Weeks
Population: A total of nine (9) participants completed both PET scans at Baseline and a follow-up scan after at least 18 weeks of treatment with RNS60 (study drug).
Measure: Mean (95% Confidence Interval); unit: Ratio
Arm/Group | RNS60
Number analyzed (Participants) | 9
Ratio | 0.02 [-0.002 to 0.042]

5. Primary Outcome: Clinical Outcome: Change in Pulmonary Function From Baseline to Week 23, Measured by Slow Vital Capacity (SVC)
Description: The vital capacity (VC) (percent of predicted normal) was determined using the slow VC method. Vital Capacity is the maximum amount of air a person can expel from the lungs after a maximum inhalation. A subject's VC depends on their age, sex and height. The value is recorded as the Week 23 minus the Baseline of percent of predicted normal.Per the protocol, the first treatment was administered on Day 0 (Baseline) and the 24th treatment was administered on Day 161 (Week 23).
Time Frame: 24 Weeks
Measure: Mean (Standard Deviation); unit: percent predicted max value
Arm/Group | RNS60
Number analyzed (Participants) | 16
percent predicted max value | -3.3 (10.16)

6. Primary Outcome: Clinical Outcome: Change in Strength From Baseline to Week 23, Measured by Accurate Test of Limb Isometric Strength (ATLIS)
Description: Accurate Test of Limb Isometric Strength (ATLIS) is a non-invasive device that allows measurements of isometric strength in 12 muscle groups of the arms and legs using a standard protocol (elbow and knee flexion and extension, grip, and dorsiflexion). Results are presented as Week 23 minus Baseline of percentages of predicted normal strength based on age, gender, height, and weight using normative data. Per the protocol, the first treatment was administered on Day 0 (Baseline) and the 24th treatment was administered on Day 161 (Week 23).
Time Frame: 24 Weeks
Measure: Mean (Standard Deviation); unit: % predicted normal strength
Arm/Group | RNS60
Number analyzed (Participants) | 16
% predicted normal strength
  ATLIS Arm Measures | -9.0 (7.19)
  ATLIS Leg Measures | -9.1 (12.91)

7. Primary Outcome: Clinical Outcome: Change in Functional Status Between Baseline and Week 23, Measured by Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R)
Description: The ALSFRS-R is a quickly administered (5 minute) ordinal rating scale used to determine a subject's assessment of their capability and independence in 12 functional activities. There are 12 questions, graded by the subject 0-4 (4 is normal). Score of 0 (worst) to 48 (best). Reflects change from Baseline to Week 23 in speech and swallowing, fine motor skills, large motor skills, and breathing. Per the protocol, the first treatment was administered on Day 0 (Baseline) and the 24th treatment was administered on Day 161 (Week 23).
Time Frame: 24 Weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | RNS60
Number analyzed (Participants) | 16
scores on a scale | -5.6 (3.96)

ADVERSE EVENTS:
Time Frame: 28 weeks
Groups:
- RNS60: RNS60: RNS60 will be administered in two ways: by intravenous (IV) infusion one day a week (infusion dose: 375ml, infused over a 40-min period) and by inhalation (the remaining 6 days a week, 4 ml/day) for 28 weeks.
Arm/Group | RNS60
All-Cause Mortality (participants affected / at risk) | 1/16
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RNS60 (N=16)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RNS60 (N=16)
Vertigo (Ear and labyrinth disorders) | 1 (2)
Conjunctival Haemorrhage (Eye disorders) | 1 (1)
Eye Irritation (Eye disorders) | 1 (1)
Vision Blurred (Eye disorders) | 1 (1)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (6)
Defaecation Urgency (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (4)
Flatulence (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (2)
Chest Pain (General disorders) | 1 (1)
Fatigue (General disorders) | 3 (6)
Feeling Abnormal (General disorders) | 1 (1)
Feeling Cold (General disorders) | 1 (1)
Feeling hot (General disorders) | 1 (1)
Implant site pain (General disorders) | 1 (1)
Infusion site bruising (General disorders) | 1 (1)
Infusion site discomfort (General disorders) | 1 (1)
Infusion site extravasation (General disorders) | 2 (2)
Infusion site pain (General disorders) | 2 (2)
Injection site bruising (General disorders) | 2 (2)
Injection site extrvasation (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (5)
Sinusitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4)
Animal bite (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 4 (7)
Fall (Injury, poisoning and procedural complications) | 11 (47)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 3 (6)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Stoma site pain (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 6 (13)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Tension headache (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Mood altered (Psychiatric disorders) | 1 (1)
Chromaturia (Renal and urinary disorders) | 1 (1)
Urine odour abnormal (Renal and urinary disorders) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (2)
Skin lesion excision (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-05): https://cdn.clinicaltrials.gov/large-docs/71/NCT02525471/Prot_SAP_000.pdf